CLINICAL TRIAL: NCT00352716
Title: Efficacy of Smecta in Combination With Oral Rehydration in the Treatment of Acute Watery Diarrhoea in Infants and Children. A Phase IIIB, Placebo, Controlled, Randomized, Double-blind, Parallel Groups, Multicenter Study.
Brief Title: Effectiveness of Smecta in the Treatment of Acute Diarrhoea in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2-31-00250-100
Record Dates: First submitted 2006-07-13; First posted 2006-07-17 (Estimated); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Diarrhoea
MeSH Terms: conditions — Diarrhea | interventions — smecta; Smectite; Duration of Therapy

INTERVENTIONS:
Drug: Smecta (Diosmectite), duration of treatment - 7 days

SUMMARY:
The purpose of this study is to evaluate the effectiveness of Smecta at decreasing stool weight, when compared to placebo, in the treatment of acute diarrhoea in children.

ELIGIBILITY:
Inclusion Criteria:

* male
* acute watery diarrhoea defined as at least 3 watery stools per 24 hours
* duration of watery diarrhoea of less than 72 hours and with at least one watery stool during the last 12 hours
* dehydration signs requiring oral rehydration according to current WHO guidelines

Exclusion Criteria:

* severe dehydration that needs IV therapy
* presence of gross blood in stools
* fever > 39 degrees Celsius
* current treatment by an antidiarrheal medication

Ages: 1 Month to 36 Months | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2006-06; Primary Completion 2007-02-01 (Actual); Study Completion 2007-02-01 (Actual)

PRIMARY OUTCOMES:
Cumulative faecal output (g/kg of body weight) | 72 hours after first study drug intake

SECONDARY OUTCOMES:
Cumulative faecal output (g) | 72 hours after first study drug intake
Faecal output (g/kg of body weight) per day | 72 hours after first study drug intake
Duration of watery diarrhoea (time of first study drug intake to watery diarrhoea disappearance) | 7 days after first study drug intake
Percentage of children withdrawn from the study due to IV rehydration (according to WHO guideline) | 7 days after first study drug intake
Percentage of body weight gain at H72 and Day 7 in comparison with body weight at inclusion | Till 7 days after the first study drug intake
Percentage of children with at least one formed stool (H12, H24, H36, H48, H60, H72, then daily until Day 7) | Till 7 days after first study drug intake
Daily until Day 7: stool frequency, watery stool number, formed stool number, soft stool number, percentage of patients with bottom skin irritation, percentage of patients with anal irritation, appetite on a 100mm visual analogue scale | Till 7 days after first study drug intake
Tolerance of Smecta (assessed via adverse event reporting) | Till 7 days after the end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (13):
- Peru (13):
  - Instituto Especializado de Salud del Niño, Breña
  - Hospital de Vitarte, Cercado
  - Hospital General de Huacho, Huacho
  - Hospital Regional de Ica, Ica
  - Hospital Nacional Hipólato Unanue, La Molina
  - Clinica San Juan Bautista, Lima
  - Clinica San Pablo Sede Norte, Lima
  - Hospital Municipal Los Olivos, Lima
  - Hospital San Bartolomé, Lima
  - Hospital San Juan de Lurigancho, Lima
  - Hospital Nacional Cayetano Heredia, San Borga
  - Hospital Nacional Daniel Alcides Carrión, San Miguel
  - Hospital Emergencias Pediátricas, Zárate